CLINICAL TRIAL: NCT06898242
Title: Early Myofascial Manual Treatment in Subjects With Spasticity Following Acquired Brain Injury
Acronym: MyosABI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, PADUA LUCA, associated professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6661
Record Dates: First submitted 2025-03-14; First posted 2025-03-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Brain Injury; Brain Injury, Vascular; Brain Injuries, Traumatic
Keywords: acquired brain injury; traumatic; spasticity; myofascial manual treatment
MeSH Terms: conditions — Brain Injuries; Cerebrovascular Trauma; Brain Injuries, Traumatic; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: rehabilitative treatment following rehabilitation project plus manual myofascial treatment (Experimental): Partecipant in group A will perform normal rehabilitative treatment as foreseen by the rehabilitation project plus manual myofascial treatment on the upper and lower limbs with a frequency of 2 times a week for a maximum of 30 minutes for 4 weeks. In particular, on the upper limbs, manual myofascial treatment will be applied in all sessions to the intraosseous membrane and if necessary to the palmar fascia, and brachial fascia sites. On the lower limbs, it will be applied in all sessions to the intraosseous membrane and if necessary to the plantar fascia, and crural fascia sites.
  Interventions: Other: Manual myofascial treatment direct to upper and lower limb; Other: Rehabilitative treatment following rehabilitation project
- Group B: rehabilitative treatment following rehabilitation project (Active Comparator): Partecipant in group B will carry out the normal rehabilitation program, as foreseen by the rehabilitation project, for a total treatment time equal to that of the treated group.
  Interventions: Other: Rehabilitative treatment following rehabilitation project

INTERVENTIONS:
Other: Manual myofascial treatment direct to upper and lower limb — Manual treatment direct specifically on fascia connective tissue
  Arms: Group A: rehabilitative treatment following rehabilitation project plus manual myofascial treatment
Other: Rehabilitative treatment following rehabilitation project — Intensive multidisciplinary rehabilitation program for at least 180 minutes/day, 6 days a week, following rehabilitation project

SUMMARY:
Spasticity is characterized by an increase in muscle tone that is velocity-dependent and caused by the exaggeration of the stretch reflex. Clinically, it is found in 70-85% of patients with spinal cord injury at one year, 40-45% in patients with stroke at 12 months, and 25% in patients with traumatic brain injury at one year.

The term 'Severe Acquired Brain Injury' refers to a condition characterized by brain damage that causes a coma with an acute phase score of 8 on the Glasgow Coma Scale (GCS), lasting more than 24 hours. It may be caused by vascular, traumatic, anoxic, infectious, toxic-metabolic, or neoplastic damage, which can cause multiple and complex sensory, cognitive, and behavioral impairments that lead to significant disability. Spasticity occurs frequently in patients with GCA, often at an early stage, with serious repercussions on the rehabilitation process and outcome.

Numerous studies indicate that spasticity due to neurological damage is supported, in addition to hyperexcitable stretch reflexes, by changes in the connective tissues of the peripheral limbs that increase muscle resistance to passive movement. After neurological damage, and starting 1 week after immobilization, alterations in the muscles and connective tissue can be observed: changes in the muscle fibers, changes in the collagen tissue, and changes in the properties of the tendons. It is believed that the quantitative and qualitative changes in the intramuscular connective tissue contribute to the deterioration of the properties and functions of the immobilized muscle, which contributes to the establishment and progression of spasticity.

In patients with spastic paresis, therapeutic interventions are intended to prevent prolonged shortening of the muscles and mobilize the affected areas. According to recent research, the connective tissue is particularly sensitive to mechanical stress, particularly deep manual manipulation and vibration. Several studies have suggested that myofascial release therapy can be a complementary treatment in patients with neurological disorders to reduce muscle spasticity and increase joint mobility.

Myofascial release techniques can be hypothesized to be a valid integrated treatment for spasticity in patients with sequelae from GCA, but their use in this area has been little studied and no studies have been conducted in the post-acute period of intensive hospitalization.

The purpose of the present study is to determine whether manual myofascial release techniques, applied to the upper and lower limbs, are safe, tolerable, and effective in modifying the degree of spasticity and improving functional activity in patients with GCA. Additionally, changes in muscle structure will be evaluated by ultrasound: cross-sectional area, anteroposterior diameter, and pennation angle.

Finally, we will measure the effects of manual myofascial treatment stimulation by measuring electrodermal activity (EDA), which is a non-invasive method in which an electrode bracelet is applied to the patient's right wrist to measure the electrical conductance of the skin, which is a function of the autonomic nervous system, which is controlled by the sweat glands. Various sensory stimulations, including visual, auditory, olfactory, tactile, vestibular, and proprioceptive stimulations, can produce a physical sensation that can influence the patient's sensorimotor output, resulting in physiological changes in the activity of the ANS as a consequence of the processing of sensory afferents. A response to an appropriate sensory stimulus can be regarded as a manifestation of a change in consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Aquired brain injuries from 40 days to 6 months after the event
* Spasticity at upper orvlower limbs quantified at MAS scale >= than 1
* Age >= 18 years
* Patient/Caregiver ability to understand and sign the informed consent

Exclusion Criteria:

* Spasticity at MAS scale > 2
* Non consolidatetd fracture and/or muscle injuries to the limbs
* Deep vein thrombosis
* Neoplasms
* Hemodynamic instability
* Local infections to the limbs
* Recent treatment with botulinum toxin (within 40 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2026-03-24 (Estimated)

PRIMARY OUTCOMES:
Modification of spasticity through Modified Ashworth Scale | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation of changes in the degree of spasticity of upper and lower limbs through Modified Ashworth Scale (lower degree 0: no increase in muscle tone; maximum degree 4: affected part rigid in flexion or extension)

SECONDARY OUTCOMES:
Tolerance and safety of treatment | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation of safety and tolerability of treatment throught Pain Assessment in Advanced Dementia scale (minimum degree 0: no pain; maximum degree 10: maximum pain)
Evaluation of changes in the degree of functional use of the upper and lower limbs through Motricity Index Scale | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Motricity Index Scale: minimum degree 0: no movement; maximum degree: movement performed with normal force

OTHER OUTCOMES:
Changes in muscle echostructure | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation in muscle echostructure through assessment of cross sectional area (Unit of Measure: cm^2) at medial gemellus muscle and biceps brachii muscle.
Changes in muscle echostructure | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation of muscle echostructure through assessment of anterior-posterior diameter (unit of measure: mm) at medial gemellus muscle and biceps brachii muscle.
Changes in muscle echostructure | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation of muscle echostructure through assessment of Heckmatt Index at medial gemellus muscle and biceps brachii muscle (unit of measure: prime numbers from 1 to 4; 1: normal aspect of muscle echostructure, clear bone echo; 4: high echointensity of muscle, absent bone echo)
Changes in muscle echostructure | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow up (T2)
  Evaluation of muscle echostructure through assessment of pennation angle at medial gemellus muscle and biceps brachii muscle (unit of measure: degrees)
Evaluation of electrodermal activity | Changes from baseline (T0), 4 weeks of treatment (T1), 4 weeks of follow-up (T2)
  Evaluation of modification of skin conductance through assessment of modification of electrodermal activity (unit of measure: prime numbers)

CONTACTS AND LOCATIONS:
Overall Officials: Luca Padua, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Neuroriabilitazione ad Alta Intensità COD. 75 Policlinico Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozcakar L, Ata AM, Kaymak B, Kara M, Kumbhare D. Ultrasound imaging for sarcopenia, spasticity and painful muscle syndromes. Curr Opin Support Palliat Care. 2018 Sep;12(3):373-381. doi: 10.1097/SPC.0000000000000354. PMID 29912727
- [Background] Posada-Quintero HF, Chon KH. Innovations in Electrodermal Activity Data Collection and Signal Processing: A Systematic Review. Sensors (Basel). 2020 Jan 15;20(2):479. doi: 10.3390/s20020479. PMID 31952141
- [Background] Heckmatt JZ, Leeman S, Dubowitz V. Ultrasound imaging in the diagnosis of muscle disease. J Pediatr. 1982 Nov;101(5):656-60. doi: 10.1016/s0022-3476(82)80286-2. PMID 7131136
- [Background] Dietz V, Sinkjaer T. Spastic movement disorder: impaired reflex function and altered muscle mechanics. Lancet Neurol. 2007 Aug;6(8):725-33. doi: 10.1016/S1474-4422(07)70193-X. PMID 17638613
- [Background] Stecco C, Day JA. The fascial manipulation technique and its biomechanical model: a guide to the human fascial system. Int J Ther Massage Bodywork. 2010 Mar 17;3(1):38-40. doi: 10.3822/ijtmb.v3i1.78. No abstract available. PMID 21589701
- [Background] Trompetto C, Marinelli L, Mori L, Pelosin E, Curra A, Molfetta L, Abbruzzese G. Pathophysiology of spasticity: implications for neurorehabilitation. Biomed Res Int. 2014;2014:354906. doi: 10.1155/2014/354906. Epub 2014 Oct 30. PMID 25530960
- [Background] Hinz B. The myofibroblast: paradigm for a mechanically active cell. J Biomech. 2010 Jan 5;43(1):146-55. doi: 10.1016/j.jbiomech.2009.09.020. Epub 2009 Oct 3. PMID 19800625
- [Background] Stecco A, Pirri C, Caro R, Raghavan P. Stiffness and echogenicity: Development of a stiffness-echogenicity matrix for clinical problem solving. Eur J Transl Myol. 2019 Sep 12;29(3):8476. doi: 10.4081/ejtm.2019.8476. eCollection 2019 Aug 2. PMID 31579488